CLINICAL TRIAL: NCT03017612
Title: A Prospective, Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of the ReVision Optics, Inc., Raindrop Near Vision Inlay for the Improvement of Near and Intermediate Vision in Pseudophakic Subjects
Brief Title: A Clinical Trial to Evaluate the Safety and Effectiveness of the Raindrop Near Vision Inlay for Pseudophakic Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of inlay from no bevel to bevel design
Sponsor: ReVision Optics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P13-0064
Record Dates: First submitted 2015-02-12; First posted 2017-01-11 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Presbyopia
Keywords: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Experimental): Evaluating the safety and effectiveness of the raindrop near vision inlay implanted in bilateral pseudophakic subjects
  Interventions: Device: Raindrop Near Vision Inlay

INTERVENTIONS:
Device: Raindrop Near Vision Inlay — A single-arm study to evaluate the effectiveness of a 2 mm corneal inlay (Raindrop Near Vision Inlay) for the treatment of presbyopia (age-related near vision loss). The anterior curvature of the cornea is re-shaped after implanting the Raindrop Near Vision Inlay in the non-dominant eye under a femtosecond laser flap to improve near and intermediate vision.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Raindrop Near Vision Inlay implanted in bilateral pseudophakes with presbyopia for improvement of near and intermediate vision. The ReVision Optics corneal inlay is a 2.0-mm, 30-micron inlay made of a hydrogel material, implanted under a lasik flap. Subjects must require reading add from +1.50 D to +2.50 D. Subjects must have a preoperative manifest refraction spherical equivalent of -0.50 to +1.00 D with no more than 0.75 D of refractive cylinder. The Raindrop Near Vision Inlay will be implanted in the non-dominant eye.

DETAILED DESCRIPTION:
Presbyopia is a natural outcome of pseudophakic subjects with monofocal or toric intraocular lenses. Treatment of pseudophakic presbyopia generally consists of reading glasses, contact lenses, or monovision LASIK, which allows the patient to see near objects. All these options suffer limitations from the patient perspective. For example, reading glasses can easily be lost or not conveniently available. Multifocal contact lenses suffer from visual symptoms and instability due to potential rotation and movement of the contact lenses on the surface of the cornea. And, successful monovision is generally limited to patients with a history of successful use of contact lenses for monovision, and even in these eyes, monovision is associated with a substantial decrease in stereo acuity and contrast sensitivity.

ReVision Optics has developed the Raindrop Near Vision Inlay for the correction of near and intermediate vision. The inlay is the same refractive index as the human cornea. The inlay is placed in the non-dominant eye, centered over the pupil after a corneal flap (LASIK) has been made. The Raindrop Near Vision Inlay is expected to provide low induction of visual symptoms and improvement of near and intermediate vision in emmetropic subjects with presbyopia. This technology may also demonstrate potential clinical utility in bilateral pseudophakic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide informed consent, have signed the written informed consent form, and been given a copy.
2. Subjects must be bilateral pseudophakic adults with presbyopia, needing reading add from +1.50 D to +2.50 D.
3. Subjects must have uncorrected near visual acuity worse than 20/40 and better than 20/200 in the non-dominant eye.
4. Subjects must have an uncorrected distance visual acuity of 20/25 or better in both eyes.
5. Subjects must have distance and near visual acuity correctable to at least 20/20 in both eyes.
6. Subjects must have a manifest refraction spherical equivalent (MRSE) between - 0.50 and +1.00 D with no more than 0.75 D of refractive cylinder in the non- dominant eye.
7. Subjects must have a tear break-up time (TBUT) of ≥8 seconds.
8. Subjects must have a central corneal thickness of between 500 and 600 microns in the non-dominant eye.
9. Subjects must have an average corneal power of ≥ 41.00 D and ≤ 47.00 D in the non-dominant eye.
10. Subjects must have a photopic pupil size of ≥3.0 mm, in the non-dominant eye.
11. Subjects must have an estimated endothelial cell count of ≥ 2000 cells/mm2 in the non-dominant eye.
12. Subjects must be willing and able to return for scheduled follow-up examinations for 24 months after surgery.
13. Subjects must have documented monovision tolerance.
14. Subjects must have a minimum of 3 months between cataract surgery and implantation of the Raindrop Near Vision Inlay in the non-dominant eye.
15. Subjects must be able to demonstrate refractive stability after cataract surgery (e.g. No change in MRSE greater than ± 0.50 D within the last 2 consecutive visits at least 2 months apart) in the non-dominant eye.
16. Subjects must have a clear or open posterior capsule in the non-dominant eye. -

Exclusion Criteria:

* 1. Subjects with anterior chamber IOLs, or posterior chamber, accommodating, or multifocal intraocular lenses (IOLs) in either eye.

  2. Subjects with anterior segment pathology in either eye.

  3. Subjects who have worn soft or rigid contact lenses within the past 30 days in the eye to be treated.

  4. Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease (e.g., meibomian gland dysfunction), or any corneal abnormality (including endothelial dystrophy, guttata, recurrent corneal erosion, etc.) in either eye.

  5. Subjects with ophthalmoscopic signs of keratoconus (or keratoconus suspect) in either eye.

  6. Subjects with distorted or unclear corneal mires on topography maps of the non- dominant eye.

  7. Subjects who require canthotomy to generate a corneal flap in the non-dominant eye.

  8. Subjects with macular degeneration, retinal detachment, or any other fundus pathology that would prevent an acceptable visual outcome in either eye.

  9. Subjects who have undergone previous corneal surgery including LASIK surgery in the non-dominant eye.

  10. Subjects with a history of herpes zoster or herpes simplex keratitis.

  11. Subjects who have a history of steroid-responsive rise in intraocular pressure, preoperative IOP > 21 mm Hg, glaucoma, or are a glaucoma suspect in either eye.

  12. Subjects with a history of uncontrolled diabetes, autoimmune disease connective tissue disease, or clinically significant atopic syndrome.

  13. Subjects on chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immunocompromised subjects.

  14. Subjects who are using ophthalmic medication(s) other than artificial tears for treatment of any ocular pathology excluding ocular allergy.

  15. Subjects using systemic medications with significant ocular side effects.

  16. Subjects with known sensitivity to planned study concomitant medications.

  17. Subjects who are participating in any other clinical trial during the course of this clinical investigation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Steinert, MD, Study Chair — Interim Dean, School of Medicine; Irving H. Leopold Professor of Ophthalmology; University of Californa, Irvine, CA
Locations (6):
- United States (6):
  - Harvard Eye Associates, Laguna Hills, California
  - Coastal Vision, Orange, California
  - Chu Vision Institute, Bloomington, Minnesota
  - Key-Whitman Eye Center, Dallas, Texas
  - Carter Eye Center, Dallas, Texas
  - Parkhurst-NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Study
Started | 13
Completed | 11
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  African American | 1
  Asian | 0
  Hispanic | 2
  Other | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Implanted Eyes With Improvement in Uncorrected Near Vision
Description: 75% of implanted eyes should achieve uncorrected near visual acuity (40cm/16in) of 20/40 or better
Time Frame: 12 months postoperatively
Measure: Number; unit: Percentage of Implanted Eyes
Arm/Group | Single Arm Study
Number analyzed (Participants) | 13
Percentage of Implanted Eyes | 100

2. Secondary Outcome: Preservation of Best Corrected Visual Acuity
Description: Fewer than 5% of eyes should lose two lines or more of best corrected distance and near visual acuity and less than 1% of eyes with preoperative best corrected visual acuity (BCVA) of 20/20 should have best corrected distance and near visual acuity worse than 20/40
Time Frame: at 6 months postoperatively and all subsequent time points up to 24 months
Measure: Number; unit: Percentage of Implanted Eyes
Arm/Group | Single Arm Study
Number analyzed (Participants) | 12
Percentage of Implanted Eyes | 92

3. Secondary Outcome: Percentage of Implanted Eyes With a Postoperative Manifest Refraction Astigmatism That Increased From Baseline by Greater Than 2.00 D
Description: Fewer than 5% of eyes should have postoperative manifest refractive astigmatism that increases from baseline by greater than 2.00 D
Time Frame: At 6 months postoperatively and all subsequent time points up to 24 months
Measure: Number; unit: Percentage of Implanted Eyes
Arm/Group | Single Arm Study
Number analyzed (Participants) | 13
Percentage of Implanted Eyes | 0

4. Secondary Outcome: Occurrence of Adverse Events
Description: Any specific adverse event should occur in less than or equal to 5% of eyes.
Time Frame: During the length of the study, up to 24 months
Measure: Number; unit: Occurrence of specific adverse events
Arm/Group | Single Arm Study
Number analyzed (Participants) | 13
Occurrence of specific adverse events
  Intraocular Pressure increase | 2
  Inlay Explant | 2
  Diffuse Lamellar Keratitis | 1
  Loss of BCVA due to late onset of haze | 1
  Hospitalization | 1
  Epiretinal Membrane | 1

5. Secondary Outcome: Uncorrected Intermediate Visual Acuity
Description: 75% of eyes should achieve uncorrected intermediate visual acuity (80 cm/32 in) of 20/40 or better
Time Frame: at 12 months postoperatively
Measure: Number; unit: Percentage of Implanted Eyes
Arm/Group | Single Arm Study
Number analyzed (Participants) | 12
Percentage of Implanted Eyes | 92

ADVERSE EVENTS:
Time Frame: 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=13)
Hospitalization due to triple arthrodesis surgery (secondary to muscular dystrophy) (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=13)
Increase in intraocular pressure > 10mmHg above baseline (Eye disorders) | 2 (2)
Inlay explant (Eye disorders) | 2 (2)
Diffuse Lamellar Keratitis (DLK) (Eye disorders) | 1 (1)
Loss of BCVA due to late onset of haze (Eye disorders) | 1 (1)
Epiretinal Membrane (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agreed to hold this information in confidence and not to disclose it to any third parties for a period of three years from the date of this agreement, or until this information becomes a matter of public knowledge or until a formal agreement for that purpose has been entered into by the parties.